CLINICAL TRIAL: NCT06238011
Title: Effect of Dexmedetomidine on Attenuation Hemodynamic Response in Coronary Artery Bypass Graft Surgical Patients: A Randomized Double Blind Controlled Trial
Brief Title: Dexmedetomidine vs Control on Attenuation Hemodynamic Response to Noxious Stimuli in CABG Surgical Patients
Acronym: CABG
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sawanpracharak hospital (Other)
Responsible Party: Principal Investigator, Padet Boonmark, Clinician at Department of Anesthesiology, Sawanpracharak hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: padetboonmark; sawanpracharakhospital (Registry Identifier: PBoonmark)
Record Dates: First submitted 2024-01-15; First posted 2024-02-02 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-02

CONDITIONS: CABG
Keywords: dexmedetomidine
MeSH Terms: interventions — Dexmedetomidine; Saline Solution

STUDY DESIGN:
Intervention Model Description: A randomized controlled trial was conduct between January2024 and March2024 at Sawanpracharak hospital, Thailand, Of 60 patients undergoing elective CABG surgery, 30 were assigned to group dexmedetomidine and 30 to group control. Dexmedetomidine prepared by nurse anesthetist in contraction 0.1mcg/kg/ml total volume 50 ml. Loading 60ml/hour in 10 minutes before induction of anesthesia then 5ml/hour until on cardiopulmonary bypass (1mcg/kg in 10 min then 0.5mcg/kg/hour). Group control received normal saline 60ml/hour in 10 minutes then 5ml/hour
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexmedetomidine (Active Comparator): Patient in this arm will receive dexmedetomidine loading 60ml/hour before induction of anesthesia then 5ml/hour until the patient on cardiopulmonary bypass
  Interventions: Drug: Dexmedetomidine
- Normal Saline (Placebo Comparator): Patient in this arm will receive normal saline loading 60ml/hour before induction of anesthesia then 5ml/hour until the patient on cardiopulmonary artery bypass
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Dexmedetomidine — Dexmedetomidine(Precedex Pfizer) prepared in concentration 0.1 mcg/kg/ml total volume50 ml by nurse anesthetist at preprocedure room, start dexmedetomidine by anesthesiologist at operating room loading 60 ml/hour for 10 minutes before induction of anesthesia then 5ml/hour until the patient on cardiopulmonary bypass (loading 1mcg/kg in 10 minutes then 0.5 mcg/kg/hour). Record patients data by nurse anesthetist
  Other Names: Precedex
  Arms: Dexmedetomidine
Drug: Normal saline — Normal Saline total volume50 ml prepared by nurse anesthetist at preprocedure room, start Normal Saline by anesthesiologist at operating room loading 60 ml/hour for 10 minutes before induction of anesthesia then 5ml/hour until the patient on cardiopulmonary bypass. Record patients data by nurse anesthetist
  Arms: Normal Saline

SUMMARY:
Aim to study efficacy of dexmedetomidine to attenuate hemodynamic response to intubation, skin incision, sternotomy and aortic cannulation

DETAILED DESCRIPTION:
A randomized controlled trial was conduct between January2024 and March2024 at Sawanpracharak hospital, Thailand. Of 60 patients undergoing elective coronary artery bypass graft, 30 were assigned to group dexmedetomidine and 30 to group control. Dexmedetomidine prepared by anesthetist nurse in concentration 0.1 microgram/kg/ml total volume 50 ml. loading dose 60 ml/hour for 10 minutes before induction of anesthesia then 5ml/hour until the patient on cardiopulmonary bypass (loading dose 1 microgram/kg for 10 minutes then 0.5 microgram/kg/hour). Group control receive normal saline 60ml/hour for 10minutes then 5 ml/hour

ELIGIBILITY:
Inclusion Criteria:

* patients schedule for CABG
* American Society of Anesthesiologist (ASA) class II-III

Exclusion Criteria:

* anticipated difficult intubation
* body mass index> 30 kg/m2
* Ejection Fraction < 40%
* left main coronary artery occlusion >50%
* left bundle branch block
* severe valvular heart disease
* severe pulmonary, renal, hepatic disease
* neurologic disease
* preoperative medication with methyldopa or clonidine

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-02-28 (Estimated); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-05-10 (Estimated)

PRIMARY OUTCOMES:
heart rate, blood pressure(systolic blood pressure, diastolic blood pressure, mean blood pressure) | during surgery
  1. heart rate in beat per minute 1.1just after loading dose 1.2 before intubation 1.3at1,3,5 minute after intubation 1.4 before skin incision 1.5 1,3,5 minutes after skin incision 1.6 before sternotomy 1.7 1,3,5 minutes after sternotomy
  2. Blood pressure (SBP, DBP,MAP)in mmHg 2.1 just after loading dose 2.2 before intubation 2.3 1,3,5 minutes after intubation 2.4 before skin incision 2.5 1,3,5 minute after skin incision 2.6 before sternotomy 2.7 1,3,5 minutes after sternotomy

SECONDARY OUTCOMES:
dose nicardipine | pre- aortic cannulation period , during surgery
  dose nicardipine in milligrams to control systolic blood pressure 80-90 mmHg at aortic cannulation period

CONTACTS AND LOCATIONS:
Overall Officials: Padet Boonmark, MD, Principal Investigator — Sawanpracharak hospital Thailand
Locations (1):
- Sawanpracharak Hospital, Nakhon Sawan, Nakhonsawan, Thailand

REFERENCES:
- [Background] Poon WH, Ling RR, Yang IX, Luo H, Kofidis T, MacLaren G, Tham C, Teoh KLK, Ramanathan K. Dexmedetomidine for adult cardiac surgery: a systematic review, meta-analysis and trial sequential analysis. Anaesthesia. 2023 Mar;78(3):371-380. doi: 10.1111/anae.15947. Epub 2022 Dec 19. PMID 36535747